CLINICAL TRIAL: NCT04208633
Title: Fellow Eye Study Evaluating Correlation Between Sulcus Anatomy and Ocular Parameters Using Ultrasound Biomicroscopy (UBM) After Horizontal or Vertical Placement of the Intraocular Lens (IOLs) in the Capsular Bag
Brief Title: Correlation Between Sulcus Anatomy and Other Parameters After Horizontal & Vertical Intraocular Lens (IOLs) Placements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 145273
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Cataract; Pseudophakia
Keywords: cataract; pseudophakia; intraocular lens; ciliary sulcus; anatomy
MeSH Terms: conditions — Cataract; Pseudophakia

STUDY DESIGN:
Intervention Model Description: Fellow eye comparison when one eye has the intraocular lens placed in horizontal and other in vertical axis.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizontal placement of the intraocular lens (Other): The eyes randomised to have horizontal placement of intraocular lenses
  Interventions: Procedure: Horizontal placement of the intraocular lens in the capsular bag
- Vertical placement of the intraocular lens (Other): Fellow eye receiving vertical placement of intraocular lens.
  Interventions: Procedure: Vertical placement of the intraocular lens in the capsular bag

INTERVENTIONS:
Procedure: Horizontal placement of the intraocular lens in the capsular bag — The eyes will be randomized (1:1) using a dedicated computer programme prior to the start of the study to have a vertical or horizontal placement of the intraocular lens in the capsular bag. The 0 and 180 degrees will be marked on the slit lamp prior to the surgery. The axes of the IOL will be orientated in reference to the midpoint of the optic haptic junction of the IOL. the fellow eye will receive the opposite placement (horizontal or vertical) of the IOL.
  Arms: Horizontal placement of the intraocular lens
Procedure: Vertical placement of the intraocular lens in the capsular bag — The eyes will be randomized (1:1) using a dedicated computer programme prior to the start of the study to have a vertical or horizontal placement of the intraocular lens in the capsular bag. The 0 and 180 degrees will be marked on the slit lamp prior to the surgery. The axes of the IOL will be orientated in reference to the midpoint of the optic haptic junction of the IOL. the fellow eye will receive the opposite placement (horizontal or vertical) of the IOL.
  Arms: Vertical placement of the intraocular lens

SUMMARY:
Usually following cataract surgery patients would expect to have normal distance vision and not require the use of distance glasses. However, in clinical practice desired vision post cataract surgery is not achieved sometimes. In such cases a piggyback lens is used to enhance the visual outcome. This lens is placed in the ciliary sulcus (space between the iris and the lens). Often this piggyback lens is not the best fit for the ciliary sulcus space and it moves. This study will be using ultrasound biomicroscopy to measure the ciliary sulcus dimensions pre and postoperatively to estimate the normal anatomy and it's variations. Patients in this study will be randomised as to which way the intraocular lens is placed in the eye (horizontally or vertically) at the time of their cataract surgery. Patients requiring cataract surgery in both eyes will be identified from the Eye Hospital at the Royal Sussex County Hospital. Patients will be in the study for up to 6 months from being identified as suitable through to the operation in the 2nd eye and a final study visit.

DETAILED DESCRIPTION:
Study Design This is a prospective, fellow eye randomised study.

Recruitment

A sample size of 92 eyes (46 patients) was calculated. Patients will be recruited at the Sussex Eye Hospital preoperative cataract assessment clinics where they will be screened and given a patient information sheet by a member of the research team if they can be recruited. They will be allowed to take this home to discuss with their family/friends and/or GP. They will be asked if the research team could contact them in a weeks time to discuss the study and the plan for the day of their surgery (which is their next NHS visit). Patients can then agree or decline to participate in the study . If they decline, their normal NHS pathway will continue. If they accept, written informed consent will be taken on the day of surgery as well as any extra imaging required. The key points of the trial will be reiterated and the patient will be invited to ask any questions. All members of the research team are NIHR GCP trained. All research patients will undergo surgery by the same surgeon and attend for post-operative follow-up at the Sussex Eye Hospital. In addition at this visit a research appointment will be made to undertake the research scans and examinations (see details below) by an experienced member of our research team. The research team including the surgeon cannot be blinded as the obvious direction of placement of the intraocular lens will be visible during surgery and during examination.

Pre-operative appointment

Consent If the patient would like to participate they will be asked to read and sign a consent form. If the patient gives consent for their GP to be notified of their participation in the study a letter will be sent to the GP.

Standard pre-operative protocol for all NHS patients:

1. Unaided and best corrected distance visual acuity
2. Intraocular pressure measurement (applanation tonometry)
3. Optical or ultrasound biometry for lens power calculation
4. Slit lamp examination of the eye (by a doctor) including dilated fundus evaluation For non-standard (research) measurements, patients will be asked to return for a separate appointment. All measurements will be performed at ambient room light (undilated pupil).

The assessment will continue as follows:

1. Scheimpflug scans (Pentacam)
2. Anaesthesia of the eye with proxymetacaine 1%
3. Measurement using digital calipers of the white-to-white diameter Carbomer gel will be applied to protect the cornea before application of ultrasound probe
4. Contact ultrasound biomicroscopy images will be taken in 4 axes: vertical, horizontal, temporal oblique and nasal oblique. The patient will be asked to fixate with the fellow eye on a target to maintain fixation and avoid accommodation. The examination will be performed with undilated pupils.

Surgery

All surgery will be carried out by the same surgeon (Principal Investigator) who is an experienced senior Ophthalmic Surgeon. This is to avoid any surgery-induced study biases. Surgery will be performed employing a standardized technique with aspheric monofocal intraocular lenses. The eyes will be randomized (1:1) using a dedicated computer programme prior to the start of the study to have a vertical or horizontal placement of the intraocular lens in the capsular bag. The 0 and 180 degrees will be marked on the slit lamp prior to the surgery. The axes of the IOL will be orientated in reference to the midpoint of the optic haptic junction of the IOL.

Non-standard (research)intervention post-operatively on the day of surgery:

Image taken with anterior segment ocular coherence tomography.

Standard post-operative protocol for all NHS patients at 4-6 weeks:

1) Unaided and best corrected distance visual acuity 2) Intraocular pressure measurement (applanation tonometry) 3) Slit lamp examination of the eye Non-standard (research) post-operative measurements for patients enrolled in this study (performed at the time convenient to patient and the research team): All measurements will be performed at ambient room light (undilated pupil).

1. Dilated retroillumination images of the IOL immediately postoperatively (ideally on the day of the surgery)
2. Scheimpflug scans (Pentacam®) at 4-6 weeks
3. Anaesthesia of the eye with proxymetacaine 1% at 4-6 weeks
4. Carbomer gel will be applied to protect the cornea before application of ultrasound probe. The patient will be asked to fixate with the fellow eye on a target to maintain fixation and avoid accommodation. This examination performed with undilated pupils at 4-6 weeks.
5. Contact ultrasound biomicroscopy images at 4-6 weeks will be taken in 4 axes: vertical, horizontal, temporal oblique and nasal oblique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataracts undergoing cataract extraction in both eye.
* Diopters of corneal astigmatism Scheimpflug imaging (Pentacam HR, Oculus, Germany)

Exclusion Criteria:

* Less than 18 years
* Significant ophthalmic co-morbidity that may affect the anatomy of the eye
* Not competent to give fully informed consent
* Unable to have surgery and attend follow up appointment at Sussex Eye Hospital, Brighton

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
Sulcus diameter versus anterior chamber dimension | 1 month
  Correlations between sulcus diameter and anterior chamber dimensions in the 4 axes pre and post operatively and also for the differences post and pre operatively.

SECONDARY OUTCOMES:
Changes in sulcus diameter in 4 axes in eyes with vertical and horizontal placement of IOLs | 1 month
  Measured on UBM
Changes in anterior chamber depth following cataract extraction | 1 month
  Measured on UBM and Pentacam
Changes in anterior chamber diameter following cataract extraction | 1 month
  Measured on UBM and Pentacam
Rotation of the IOL in degrees from it's primary placement at 4-6 weeks at postoperative follow up. | 1 month
  Measured on retro-illumination photographs
To explore any relationship between demographics in relation to sulcus anatomy | 1 month
  Analysed from the demographics

CONTACTS AND LOCATIONS:
Overall Officials: Mayank Nanavaty, Study Chair — Brighton and Sussex University Hospitals NHS Trust
Locations (1):
- Brighton & Sussex University Hospitals NHS Trust, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nanavaty MA, Offer C, Kier C, Way C, Frattaroli P, Bremner S. Changes in the sulcus and anterior chamber after horizontal or vertical intraocular lens orientation: prospective randomized study. J Cataract Refract Surg. 2025 Nov 1;51(11):1011-1018. doi: 10.1097/j.jcrs.0000000000001727. PMID 40601404
- See also: Health Research Authority UK — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/sulcus-anatomy-using-ultrasound-biomicroscopy/